CLINICAL TRIAL: NCT07157761
Title: The Effectiveness of a Dutch Program in Preventing Criminal Exploitation: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Dutch Program in Preventing Criminal Exploitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Collaborators: VU University of Amsterdam (Other); Netherlands Institute for the Study of Crime and Law Enforcement (NSCR) (Unknown)
Responsible Party: Principal Investigator, Marit van de Mheen, PhD candidate, Utrecht University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1434.201.001.a
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Delinquency; Externalizing Behavior
Keywords: criminal exploitation

STUDY DESIGN:
Intervention Model Description: A cluster RCT will be used to determine the effectiveness of the program. Within each school, classes will be randomly assigned to either the experimental group, in which the program starts as soon as possible, or to a waitlist control group, which starts after the follow-up period (six months). Randomization to either the experimental or control group will take place using a computerized randomization in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The program is taught by a trusted teacher of the students (for example, their mentor). The program consists of a lesson of about one hour. It includes a short film and an interactive chat box that allows students to chat with the main character of the film. In addition, there is a guideline for discussing the topic in the classroom and information on where to find help.
  Interventions: Behavioral: Buit in de klas
- control group (No Intervention): This group will not participate in the program. They will receive the program afterwards, once data collection is finished.

INTERVENTIONS:
Behavioral: Buit in de klas — The program is taught by a trusted teacher of the students (for example, their mentor). The program consists of a lesson of about one hour. It includes a short film and an interactive chat box that allows students to chat with the main character of the film. In addition, there is a guideline for discussing the topic in the classroom and information on where to find help.
  Arms: experimental group

SUMMARY:
The purpose of this study is to investigate whether the prevention program 'Buit in de Klas' is effective.

DETAILED DESCRIPTION:
Due to the growing concerns about youth involvement in crime, the Dutch Government has recently provided substantial financial support to municipalities to prevent and address youth crime (Veiligheid, 2024). These funds are intended, in part, for prevention and intervention programs aimed at reducing or preventing criminal involvement among young people. Aim of this study is to examine the effectives of the prevention program "Buit in de klas". Buit in de klas is a school-based prevention program for students aged 12-20) to prevent criminal exploitation. The program is offered at secondary schools, consisting of a film and an accompanying lesson, usually as part of lessons in citizenship. The prevention program aims to empower students to protect themselves and peers from criminal exploitation (Noord Holland Samen Veilig & Garage2020., 2022).

To achieve these goals, the program has three intermediary objectives. First, it aims to improve students' knowledge to recognize early signs of risk for becoming a victim of criminal exploitation. Second, the program seeks to increase awareness of the consequences of criminal exploitation and thereby to influence cognitions and foster more negative attitudes toward criminal exploitation. Finally, the primary objective of the program is to teach students help-seeking skills when they or their peers are at risk of criminal exploitation.

The study hypothesis is that the prevention program Buit in de klas is effective in preventing criminal exploitation by increasing knowledge about the signs and consequences of criminal exploitation, enhancing empathy for children who are victims of criminal exploitation, and strengthening students' help-seeking skills.

ELIGIBILITY:
Inclusion Criteria:

* The participant is between 12-20 years old.
* The particpant attend school.

Every student who meets the inclusion criteria for the intervention program can participate in the study

Exclusion Criteria:

* Participants are younger than 12 years old or older than 20 years old.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge about criminal exploitation | baseline (T0), three months after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 6 months post-program (T2).
  Knowledge of criminal exploitation will be assessed using six questions. First, participants are asked: 'Do you know what criminal exploitation is?' Those who respond with 'yes' or 'a little' are then invited to describe, in their own words, what it entails. In addition, a multiple-choice question asks participants to select the definition that best fits criminal exploitation. A subsequent item asks: 'How well do you think you can recognize signs of criminal exploitation?' Another question assesses whether participants know someone who has been asked to engage in criminal activity, and, if so, how they recognized this.
Attitudes toward criminal exploitation | baseline (T0), three months after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 6 months post-program (T2).
  Attitudes will be measured using a questionnaire adapted from the Attitude Towards Delinquent Behaviour Questionnaire (ATDS; Menard & Huizinga, 1994). Nine items will be rated on a 4-point Likert scale, with response options ranging from 'not wrong at all' to 'very wrong.' An example item is: 'What do you think about someone your age stealing something worth more than 50 euros?. Empathy towards peers will be measured using three statements (e.g., 'I feel sorry for classmates who are treated unfairly').
Help-seeking behaviour | baseline (T0), three months after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 6 months post-program (T2).
  Will be measured using the 12-item Multidimensional Scale of Perceived Social Support (MSPSS) (Zimet et al., 1990).
  Participants rate statements such as "I have a special person who is a real source of comfort to me" and "I can talk about my problems with my family" on a 5-point Likert scale (1 = very strongly disagree to 5 = very strongly agree).
  Higher scores indicate greater levels of experienced support. And a question that assesses whether they know where to find help, either for themselves or for a peer who may be at risk of criminal exploitation.

SECONDARY OUTCOMES:
Externalizing behaviour | Baseline (T0) and 6 months after the program (T2)
  will be measured using the externalizing behavior and delinquency subscales of the Youth Self-Report (YSR) (Verhulst & Van der Ende, 1992). The instrument focuses on various externalizing behaviors, including aggression and delinquent behavior. The YSR includes items such as "I fight a lot", which are rated on a 3-point Likert scale ranging from 0 (never) to 2 (often). Higher scores on the YSR externalizing subscale indicate greater levels of externalizing behavior.

OTHER OUTCOMES:
Demographic, personal, socioeconomic, and family background | Baseline (T0)
  will be assessed through a questionnaire covering demographic information, including age, gender, ethnic identity, family composition, and financial situation (e.g., "Do you worry whether there is enough money at home?").
Parent-child relationship | baseline (T0) and at 6 months post-program (T2)
  will be assessed using statements based on the Parental Monitoring Questionnaire (Stattin & Kerr, 2000) containing three subscales: parental control, parental solicitation, and parental disclosure. Parental control contains five item, indicating the extent to which parents seek to regulate their child's behavior by requiring permission for leisure activities. Parental solicitation (five items) captures the degree to which parents proactively seek information about their child's leisure activities. Parental disclosure (5 items) reflects how openly juveniles voluntarily share such information with their parents. All items are rated on a 5-point Likert scale 1 (never) to 5 (always). Parental responsivity will be assessed using the eight-item Responsivity subscale of the Nijmegen Parenting Questionnaire (Gerris, 1993).
  Items are rated on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree).
Presence of Deviant peers | baseline (T0) and at 6 months post-program (T2)
  will be measured using the Deviant Peers Scale from the Basic Questionnaire on Peer Relationships (Weerman & Smeenk, 2005). The five -items questionnaire assesses the extent to which juveniles have deviant friends. (e.g., ''How many of your friends have robbed someone by threatening with a weapon or violence, or by using violence?'').
  Responses are given on a four-point scale (none, some, most, all). Internal consistency in previous studies was high.
  Higher scores on this scale indicate that juveniles have more deviant friends.
Problems and help-seeking | baseline (T0) and at 6 months post-program (T2)
  will be measured using a short questionnaire that has also been used in the study of Tollenaar and colleagues (Tollenaar et al., 2024). This questionnaire asks about various issues pupils may have experienced in the past six months (e.g., family problems, financial problems, or mental health issues). Respondents can indicate whether they have had any of these problems and, if so, whether they sought help and from whom (e.g., social worker, youth services, school mentor, or parents). Responses are given as yes/no options for each category, and additional openended fields allow participants to specify other sources of help or problems they experienced.
School performance | baseline (T0) and at 6 months post-program (T2)
  will be measured using an adapted version the Family, Friends, and Self (FSS) questionnaire (Simpson & McBride, 1992). The questionnaire contains five items (e.g., "How did your schoolwork go last week?"). Responses are given on a five-point scale ranging from 1 (really bad) to 5 (really good), with higher scores indicating better school performance.
  The internal consistency is good (α = .79) (Duari & Mohapatra, 2021; Simpson & McBride, 1992). Participants are also asked whom they can ask for help with their homework and whether they skip school.
Leisure time activities | baseline (T0) and at 6 months post-program (T2)
  will be assessed using a questionnaire based on the Dutch Monitor of Self-Reported Delinquency (Tollenaar et al., 2024). Participants answered two questions about where they usually spend their time after school on weekdays (Monday to Thursday) and during the weekend (Friday to Sunday). Eleven response options were provided, allowing multiple answers. Examples include going out with parents; attending a sports club; being at friends' homes; hanging out on the street with friends; or never going out/mostly staying at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Asscher, PhD., Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data can be shared in anonymized form upon request.
Supporting Information: Study Protocol
Time Frame: The data will become available after the completion of the program and data collection.